CLINICAL TRIAL: NCT04112771
Title: Effects of Penehyclidine on Postoperative Nausea and Vomiting in Patients Underging Bimaxillary Surgery: A Retrospective Cohort Study
Brief Title: Penehyclidine and Postoperative Nausea and Vomiting After Bimaxillary Surgery
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Hospital of Stomatology (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anaesthesiology and Critical Care Medicine, Peking University First Hospital
Other Study IDs: 201947098
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Penehyclidine; Postoperative Nausea and Vomiting; Bimaxillar Surgery
Keywords: Penehyclidine; Postoperative nausea and vomiting; Bimaxillary surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — penehyclidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Penehyclidine group: Penehyclindine hydrochloride was administered before anesthesia induction.
  Interventions: Drug: Penehyclidine hydrochloride
- Placebo group: Penehyclindine hydrochloride was not administered before anesthesia induction.
  Interventions: Other: No penehyclidine hydrochloride

INTERVENTIONS:
Drug: Penehyclidine hydrochloride — Penehyclidine hydrochloride was administered before anesthesia induction.
  Groups: Penehyclidine group
Other: No penehyclidine hydrochloride — Penehyclidine hydrochloride was not administered before anesthesia induction.
  Groups: Placebo group

SUMMARY:
Postoperative nausea and vomiting (PONV) are common complications after surgery. Patients undergoing orthognathic surgery are reported to have a high rate of PONV, especially those undergoing bimaxillary surgery. Activation of cholinergic system plays an important role in the development of PONV. Penehyclidine is an muscarinic antagonists which selectively block M1 and M3 receptors and is commonly used to decrease oral secretion. The purpose of this retrospective cohort study is to investigate whether use of penehyclidine is associated with a reduced risk of PONV in patients undergoing bimaxillary surgery.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) are one of the most frequent complications after surgery, and are associated with patients' dissatisfaction after anesthesia and surgery. Orthognathic surgery is widely performed for the correction of dentofacial deformities. PONV is common after orthognathic surgery. Despite of improved anti-emetic prophylaxis, patients undergoing orthognathic surgery are reported to have a high incidence of PONV, especially those after bimaxillary surgery.

It is known that activation of central cholinergic system plays an important role in the development of PONV. Muscarinic antagonists such as scopolamine can block muscarinic receptors in the cerebral cortex and produce anti-emetic effects. Penehyclidine is a new muscarinic antagonists which selectively block M1 and M3 receptors. It has fewer adverse effects compared with other anticholinergics. The purpose of this retrospective cohort study is to investigate whether use of penehyclidine is associated with a reduce risk of PONV in patients undergoing bimaxillary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years;
* Underwent elective bimaxillary surgery under general anesthesia.

Exclusion Criteria:

* Age <16 years;
* Missing data.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent bimaxillary surgery between April 1, 2018 and September 30, 2019 in Peking University Hospital of Stomatology.
Sampling Method: Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting (PONV) within 48 hours after bimaxillary surgery. | Up to 48 hours after surgery.
  Nausea was assessed by direct questioning. Vomiting was diagnosed when patients retched or expulsed intra-gastric contents.

SECONDARY OUTCOMES:
Daily prevalence of PONV. | Up to 48 hours after surgery.
  Daily prevalence of PONV on the day of surgery, as well as the first and second day after surgery.
Postoperative agitation after bimaxillary surgery. | Up to 8:00 am on the first day after surgery.
  Postoperative agitation was diagnosed when a Richmond Agitation-Sedation Scale (scale ranges from -5 to +4, with higher scale indicating severe agitation) reached +2 or more at any time within 2 hours after extubation.
Postoperative pain after bimaxillary surgery. | Up to 2 days after surgery.
  Postoperative pain was assessed with the Numeric Rating Scale (an 11-point scale where 0=no pain and 10=the worst pain). A score of 4 or more is defined a moderate-to-severe pain.
Postoperative complications during hospital stay after surgery. | Up to 30 days after surgery.
  Postoperative complications were generally defined as new-onset medical events that were harmful for patients' recovery and required therapeutic intervention.
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
In-hospital mortality after surgery. | Up to 30 days after surgery.
  In-hospital mortality after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University Hospital of Stomatology, Beijing, Beijing Municipality
  - Peking University Hospital of Stomatology, Beijing, Haidian

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myles PS, Williams DL, Hendrata M, Anderson H, Weeks AM. Patient satisfaction after anaesthesia and surgery: results of a prospective survey of 10,811 patients. Br J Anaesth. 2000 Jan;84(1):6-10. doi: 10.1093/oxfordjournals.bja.a013383. PMID 10740539
- [Background] Naran S, Steinbacher DM, Taylor JA. Current Concepts in Orthognathic Surgery. Plast Reconstr Surg. 2018 Jun;141(6):925e-936e. doi: 10.1097/PRS.0000000000004438. PMID 29794714
- [Background] Laskin DM, Carrico CK, Wood J. Predicting postoperative nausea and vomiting in patients undergoing oral and maxillofacial surgery. Int J Oral Maxillofac Surg. 2020 Jan;49(1):22-27. doi: 10.1016/j.ijom.2019.06.016. Epub 2019 Jun 21. PMID 31230771
- [Background] Phillips C, Brookes CD, Rich J, Arbon J, Turvey TA. Postoperative nausea and vomiting following orthognathic surgery. Int J Oral Maxillofac Surg. 2015 Jun;44(6):745-51. doi: 10.1016/j.ijom.2015.01.006. Epub 2015 Feb 2. PMID 25655765
- [Background] Dobbeleir M, De Coster J, Coucke W, Politis C. Postoperative nausea and vomiting after oral and maxillofacial surgery: a prospective study. Int J Oral Maxillofac Surg. 2018 Jun;47(6):721-725. doi: 10.1016/j.ijom.2017.11.018. Epub 2018 Jan 1. PMID 29301675
- [Background] Shaikh SI, Nagarekha D, Hegade G, Marutheesh M. Postoperative nausea and vomiting: A simple yet complex problem. Anesth Essays Res. 2016 Sep-Dec;10(3):388-396. doi: 10.4103/0259-1162.179310. PMID 27746521
- [Background] Han XY, Liu H, Liu CH, Wu B, Chen LF, Zhong BH, Liu KL. Synthesis of the optical isomers of a new anticholinergic drug, penehyclidine hydrochloride (8018). Bioorg Med Chem Lett. 2005 Apr 15;15(8):1979-82. doi: 10.1016/j.bmcl.2005.02.071. PMID 15808451